CLINICAL TRIAL: NCT03194763
Title: Observational Study for Feasibility and Performance of Sub-millisievert Coronary Computed Tomography Angiography (CCTA) for Coronary Artery Anomalies (CAA) in Paediatric Patients
Acronym: COROPEDIA
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: 9785
Record Dates: First submitted 2017-06-19; First posted 2017-06-21 (Actual); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Coronary Artery Anomaly, Congenital
MeSH Terms: interventions — Coronary Angiography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: coronary angiography — computed tomography acquisitions performed on a revolution CT

SUMMARY:
Congenital heart defects are the most frequent manifestation of congenital diseases (8 per 1000 live births). Imaging modalities play an increasing role in their diagnosis, follow-up, and pre/post-surgery check-up. Echocardiography usually provides a first line diagnosis, but Coronary CT Angiography (CCTA) also demonstrated its usefulness whenever accurate modelling of anatomic structures is required.

CCTA is well defined for adult patients. This is not the case for paediatric population, which rises two main difficulties:

* The use of ionising radiation in young subjects involves a very radio-sensitive population, potentially subject to multiple exams during their follow up.
* Technical issues related to young patients: No breath-holding, uncontrolled movements during acquisition, very high heart rates (making ECG gating more complex) and very small structures.

These conditions usually result in a deteriorated image quality or in radiation dose increase (retrospective gating). These two outcomes are not acceptable for both, clinician and patient.

In this study, investigators make the hypothesis that despite difficult conditions stated above, ultra-low dose acquisitions may results in diagnostic quality acquisition, thanks to state of art CT technologies combined with acquisition parameters specially designed for that purpose.

Investigators aim to demonstrate feasibility and performances of such exams.

DETAILED DESCRIPTION:
Fifty paediatric patients are to be enrolled in this study. All these patients were prescribed a coronary angiography CT as part of their follow up for a known or suspected coronary artery anomaly.

Computed Tomography acquisitions are performed on a Revolution CT (GE Healthcare) using a wide detector aperture (160 mm), last generation of iterative reconstruction algorithm and specific reconstruction software reducing cardiac motion artefacts. A rotation time of 0.28 sec is used, with a slice thickness of 0.625 mm and a 0.625 mm reconstruction interval. The acquisition is ECG-gated (prospective) with kV and mAs depending on BMI, heart rate and heart rate variability of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients from 0 to 18 years old
* Known or suspected coronary artery anomalies
* CCTA prescribed for regular follow up of the pathology
* No-objection of parents/legal representative of the patient
* Covered by social security

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients from 0 to 18 years old with known or suspected coronay artery anomalies
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
CT diagnostic performance evaluation | first day
  CT diagnostic performance evaluation using a semi-quantitative likert scale

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric and Congenital Cardiology and Pulmonology Department, Arnaud De Villeneuve University Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Le Roy J, Vernhet Kovacsik H, Zarqane H, Vincenti M, Abassi H, Lavastre K, Mura T, Lacampagne A, Amedro P. Submillisievert Multiphasic Coronary Computed Tomography Angiography for Pediatric Patients With Congenital Heart Diseases. Circ Cardiovasc Imaging. 2019 Feb;12(2):e008348. doi: 10.1161/CIRCIMAGING.118.008348. PMID 30704282